CLINICAL TRIAL: NCT04677582
Title: Vidas Activas, famiLias saludablEs (Active Lives, Healthy Families) (VALÉ)
Brief Title: VALÉ: A Multidisciplinary Childhood Obesity Treatment Program for Latino Communities
Acronym: VALÉ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117702
Record Dates: First submitted 2018-08-09; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The intervention group will receive weekly education sessions about nutrition, exercise, and behavioral health.
  Interventions: Behavioral: Vidas Activas, famiLias saludablEs (VALE)

INTERVENTIONS:
Behavioral: Vidas Activas, famiLias saludablEs (VALE) — Families and Children allocated to the intervention will receive weekly group-based meetings over a 10-week period consisting of education and activities on healthy lifestyles. Graduate students/Research Assistants trained in nutrition, exercise and clinical psychology will lead the meetings. All activities will be culturally relevant (i.e. cooking healthy Latino recipes) and Spanish speaking students will be recruited to deliver the intervention. Participants will be involved on deciding activities and projects and while some sessions will meet as a family group with parents/guardians, others will meet separately.

SUMMARY:
This proposal aims to test the initial feasibility and efficacy of a 10-week multidisciplinary pediatric weight management program among low-income Latino children, aged 5 to 11 years, from the Woodbridge, VA area. The following specific aims will be tested:

DETAILED DESCRIPTION:
Specific Aim 1: To test the acceptability of a multidisciplinary group intervention targeted towards low-income Latino families with a child who is obese.

Specific Aim 2: To test the effectiveness of the intervention by determining differences in behavioral changes (i.e. nutrition and physical activity habits), anthropometric (BMI-for-age, body fat) and clinical health outcomes (i.e. blood pressure, blood biomarkers) between children exposed to the intervention program vs. control children.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pubertal (girls must not have started menses)
* Of Latino/Hispanic descent (parent self-identified)
* BMI for age >85th percentile (based on CDC growth reference)
* Child between 5-11 years old
* Healthy (no known chronic diseases or regular medication)
* Parent/adult caregivers willing to participate in all study visits

Exclusion Criteria:

* Not of Latino/Hispanic descent
* <5 years old or >11 years old
* BMI for age <85th percentile
* Not pre-pubertal (girls have experienced their first menses)
* Child has learning deficits or acute/chronic medical condition
* Parent/guardian has no transportation or unable to participate in sessions

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline BMI at 3 months and 6 months | Baseline, 3 and 6 months
  body weight (kg)/height(m^2)
Change from Baseline Body Fat Percentage at 3 months and 6 months | Baseline, 3 and 6 months
  % via bioelectric impedance
Change from Baseline Blood Pressure at 3 months and 6 months | Baseline, 3 and 6 months
  Systolic & Diastolic Blood Pressure
Change from Baseline Waist Circumference at 3 months and 6 months | Baseline, 3 and 6 months
  cm
Change from Baseline HbA1c at 3 months and 6 months | Baseline, 3 and 6 months
  HbA1c (%)
Change from Baseline Glucose at 3 months and 6 months | Baseline, 3 and 6 months
  Glucose (mg/dL)
Change from Baseline Blood Lipids at 3 months and 6 months | Baseline, 3 and 6 months
  LDL, HDL, TRG, TC (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Jones, PhD, CSCS*D, Principal Investigator — George Mason University
Locations (2):
- United States (2):
  - Featherstone Elementary School, Woodbridge, Virginia
  - Kilby Elementary School, Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: No